CLINICAL TRIAL: NCT06734195
Title: Comparing the Synergistic Effect of Caudal Dexmedetomidine and Propofol Versus Caudal Dexmedetomidine Only or Propofol Only in Prevention of Sevoflurane Related Emergence Agitation in Pediatric Patients Undergoing Congenital Inguinal Hernia Repair: Randomized Double-blind Controlled Study
Brief Title: Comparing the Synergistic Effect of Caudal Dexmedetomidine and Propofol Versus Caudal Dexmedetomidine Only or Propofol Only in Prevention of Sevoflurane Related Emergence Agitation in Pediatric Patients Undergoing Congenital Inguinal Hernia Repair
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abudaif Abdelrazzak Abudaif eid, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sevoflurane gitation
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Sevoflurane Agitiion in Pediatric
Keywords: sevoflurane; Dexmedetomidine; Propofol
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (propofol group) (Experimental): 30 patients will receive propofol 1mg/kg before the start of skin closure, administered over 10 minutes and caudal block using 1 ml/kg of bupivacaine 0. 25 % plus 2 ml normal saline.
  Interventions: Drug: Propofol alone
- Group B (caudal dexmedetomidine group) (Experimental): 30 patients will receive caudal dexmedetomidine block using 1 ml/kg of bupivacaine 0. 25 % mixed with dexmedetomidie 1mic/kg diluted in 2 ml normal saline.
  Interventions: Drug: Dexmedetomidine
- Group C (propofol with caudal dexmedetomidine group) (Experimental): 30 patients will receive both propofol .5 mg/kg before the start of skin closure, administered over 10 minutes and caudal dexmedetomidine block using 1 ml/kg of bupivacaine 0. 25 % mixed with dexmedetomidie 1mic/kg diluted in 2 ml normal saline.
  Interventions: Drug: dexmedetomidine + propofol

INTERVENTIONS:
Drug: dexmedetomidine + propofol — Comparison of caudal dexmedetomidine + propofol sevoflurane-related emergence agitation in children undergoing congenital hernia repair.
  Arms: Group C (propofol with caudal dexmedetomidine group)
Drug: Propofol alone — 30 patients will receive propofol 1mg/kg before the start of skin closure, administered over 10 minutes and caudal block using 1 ml/kg of bupivacaine 0. 25 % plus 2 ml normal saline.
  Arms: Group A (propofol group)
Drug: Dexmedetomidine — patients will receive caudal dexmedetomidine block using 1 ml/kg of bupivacaine 0. 25 % mixed with dexmedetomidie 1mic/kg diluted in 2 ml normal saline
  Arms: Group B (caudal dexmedetomidine group)

SUMMARY:
evaluate the synergistic efficacy of propofol and caudal dexmedetomidine for postoperative EA in pediatrics aged from to 2 to 5 years maintained on sevoflurane inhalational anesthesia and scheduled for conginital inguinal hernia repair surgeries

DETAILED DESCRIPTION:
Eligibility and type of the study: This prospective randomized placebo-controlled double-blind study will be conducted after approval from the Institutional Ethics Committee and obtaining written informed consent from parents of children scheduled for conginital inguinal hernia repair procedures under general anesthesia. This study will be conducted at pediatric surgery operating theatre, Assiut University Hospitals.

Sample size:

Drugs coding and Randomization: Patients will be randomly allocated into three equal groups with the help of a computer-generated table of random numbers to receive the study drugs. One anesthesiologist, not involved in the study procedure or data collection, will prepare the study drugs in identical coded syringes. Access to these codes will be only available to one anesthesiologist who will prepare the syringes according to the study drugs used. To ensure double-blinding, the anesthetic technique and outcome data will be collected by an anesthesiologist not included in preparing study drugs or envelops coding. Also the parents will be blinded to the drug grouping of their children.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-7 years
* Both genders
* American society of anesthesiologists (ASA) physical state I-II
* Children undergoing sub-umbilical abdominal surgeries

Exclusion Criteria:

* Guardians refusal
* Congenital anomalies at the lower spine or meninges
* Increased intracranial pressure
* Skin infection at the site of injection
* Bleeding diathesis
* Known allergy to any drugs used in this study
* Children with behavioral changes; physical or developmental delay; neurological disorder or psychological disorder.
* Children on sedative or anticonvulsant medication.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2027-04-10 (Estimated); Study Completion 2028-05-10 (Estimated)

PRIMARY OUTCOMES:
postoperative EA | 24 hours
  The incidence of postoperative emergence agitation in the study groups will be evaluated by using the (PAED Score)

OTHER OUTCOMES:
Secondary outcome | baseline
  will include the study effects on: Hemodynamic parameters, Postoperative pain, Postoperative sedation, Time to the first dose of analgesia postoperatively, Total amount of rescue analgesia in first 24 h postoperatively, Complications, and Parents' satisfaction score.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Sied Abd El rahem, PROF, Study Chair — Assiut University; Sara Mohamed Mansour Fathy, DR, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore AD, Anghelescu DL. Emergence Delirium in Pediatric Anesthesia. Paediatr Drugs. 2017 Feb;19(1):11-20. doi: 10.1007/s40272-016-0201-5. PMID 27798810
- [Background] Mohkamkar M Bs, Farhoudi F Md, Alam-Sahebpour A Md, Mousavi SA Md, Khani S PhD, Shahmohammadi S BSc. Postanesthetic Emergence Agitation in Pediatric Patients under General Anesthesia. Iran J Pediatr. 2014 Apr;24(2):184-90. PMID 25535538
- [Background] Cao JL, Pei YP, Wei JQ, Zhang YY. Effects of intraoperative dexmedetomidine with intravenous anesthesia on postoperative emergence agitation/delirium in pediatric patients undergoing tonsillectomy with or without adenoidectomy: A CONSORT-prospective, randomized, controlled clinical trial. Medicine (Baltimore). 2016 Dec;95(49):e5566. doi: 10.1097/MD.0000000000005566. PMID 27930564
- [Background] Kanaya A. Emergence agitation in children: risk factors, prevention, and treatment. J Anesth. 2016 Apr;30(2):261-7. doi: 10.1007/s00540-015-2098-5. Epub 2015 Nov 24. PMID 26601849
- [Background] Brioni JD, Varughese S, Ahmed R, Bein B. A clinical review of inhalation anesthesia with sevoflurane: from early research to emerging topics. J Anesth. 2017 Oct;31(5):764-778. doi: 10.1007/s00540-017-2375-6. Epub 2017 Jun 5. PMID 28585095
- [Background] Cravero J, Surgenor S, Whalen K. Emergence agitation in paediatric patients after sevoflurane anaesthesia and no surgery: a comparison with halothane. Paediatr Anaesth. 2000;10(4):419-24. doi: 10.1046/j.1460-9592.2000.00560.x. PMID 10886700
- [Background] Feng Z, Shi X, Yan X, Zhu Y, Gu J, Zhu H, Yu W, Zhang S. Comparing the effects of dexmedetomidine versus propofol on the treatment of emergence agitation in adult patients after general anesthesia: study protocol for a randomized, superiority, controlled trial (DP-TEA Trial). Trials. 2021 Nov 16;22(1):811. doi: 10.1186/s13063-021-05743-2. PMID 34784941
- [Background] Ecoffey C. Safety in pediatric regional anesthesia. Paediatr Anaesth. 2012 Jan;22(1):25-30. doi: 10.1111/j.1460-9592.2011.03705.x. Epub 2011 Sep 20. PMID 21933301
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Background] Turkyilmaz N, Gurkan Y, Cesur S, Kus A, Solak M. [Ultrasound-guided penile nerve block for pediatric hypospadias surgery]. Agri. 2018 Apr;30(2):97-98. doi: 10.5505/agri.2016.70446. Turkish. PMID 29738062
- [Background] Yeap E, Pacilli M, Nataraja RM. Inguinal hernias in children. Aust J Gen Pract. 2020 Jan-Feb;49(1-2):38-43. doi: 10.31128/AJGP-08-19-5037. PMID 32008266
- See also: Related Info — https://www.wiley.com/en-us/Jones'+Clinical+Paediatric+Surgery%2C+7th+Edition-p-9781118777312
- See also: Related Info — https://scholar.google.co.in/citations?user=cKvhjAoAAAAJ&hl=en